CLINICAL TRIAL: NCT01905202
Title: Phase 1 Safety and Tolerability of Secretrol in Patients With Barrett's Esophagus
Brief Title: The Safety and Tolerability of Secretrol in Patients With Barrett's Esophagus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Effexus Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP404
Record Dates: First submitted 2013-07-17; First posted 2013-07-23 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Barrett's Esophagus
Keywords: Proton Pump Inhibitor; Safety; Tolerability; pH control; Bile Acid
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Secretrol (Experimental): Secretrol Capsules 80/80 once daily for 6 months
  Interventions: Drug: Secretrol

INTERVENTIONS:
Drug: Secretrol

SUMMARY:
Secretrol administered over a 6 month period to patients with Barrett's Esophagus will be safe and well tolerated. Further, pH control will be evaluated in the distal esophageal mucosa and just below the squamocolumnar junction.

DETAILED DESCRIPTION:
A majority of patients with Barrett's esophagus have poor distal esophageal pH control. Such patients frequently receive more than one dose of PPI per day in an attempt to improve esophageal pH control. Nocturnal pH control is notably difficult to achieve in many patients suffering from Barrett's esophagus. Recently, adverse effects have been associated with prolonged PPI use (defined as 1 year or longer). These include hypomagnesemia, bone fractures, Clostridium difficile induced diarrhea. High dose PPI as well as very high dose PPI usage (such as that used in hypersecretory conditions) has generally not been found to produce a different side effect or tolerability profile in humans. This study will evaluate the effects of Secretrol on tolerability, adverse effects and pH control of the distal esophagus and just below the squamocolumnar junction.

ELIGIBILITY:
Inclusion Criteria:

* Barrett's esophagus with histological confirmed Barrett's ≥ 2 cm in length and negative or indefinite for dysplasia/neoplasia.
* Ages 18 and older.
* Patients who have signed an Informed Consent Form and Health Insurance Portability and Accountability Act (HIPAA) Authorization Form.

Exclusion Criteria:

* Clinically relevant data suggesting an unknown disease and requiring further evaluation by the Primary Investigator.
* If you have a pacemaker, cardiac defibrillator or neurostimulator.
* Patients with renal failure or organ transplants.
* Patients who have known allergic reactions to Proton Pump Inhibitors.
* Participation in another study within 30 days prior to screening.
* Previous enrollment into the current study.
* Patient is the Investigator, his family member or employee at the investigational site.
* Patient known or suspected to be involved in alcohol or drug abuse.
* Known or suspected history of non-compliance with medications.
* Inability to follow the procedures of the study (e.g., due to language problems, psychological disorders)
* Patients receiving prohibited concomitant medications including PPIs, H2 blockers, sucralfate, misoprostil. Note: patient to take dose of "usual" PPI medication in morning of visit 2 and continue for the next 24 hours. After that no PPI is permitted (except Secretrol)
* Patients receiving prohibited concomitant medications including theophylline, clopidogrel, ketoconazole, digoxin, diazepam, warfarin, phenytoin, emtricitabine/nelfinavir/tenofovir, atazanavir, citalopram, emtricitabine/rilpivirine/tenofovir, rilpivirine, nelfinavir, tricyclic antidepressants, baclofen, tacrolimus, cyclosporine, cilostazol, disulfiram, methotrexate, voriconazole.
* Pregnancy or intention to become pregnant during the course of study, breast feeding, or unwillingness to use a highly effective means of contraception (oral contraception or intrauterine device).
* Unable to complete 48-hr esophageal pH monitoring.
* Prescription NSAID use or aspirin use greater than 325mg daily.
* History of upper gastrointestinal surgery, Zollinger-Ellison syndrome, esophageal stricture, peptic stricture, duodenal and ⁄ or gastric ulcer, esophageal motility disorders, IBD, AIDS, pancreatitis, malabsorption, severe cardiovascular or pulmonary disease, liver disease, active malignant disease, scleroderma, autonomic or peripheral neuropathy, myopathy, any underlying disease or medication that might affect the lower esophageal sphincter pressure or increase the acid clearance time.
* Were unable or unwilling to fully complete all stages of the study.
* Unable to sign informed consent or inability to give fully informed consent due to language problems, psychological disorder or mental deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | at 6 months

SECONDARY OUTCOMES:
Number of participants who develop C. difficile induced diarrhea | Over 6 months

OTHER OUTCOMES:
Gastrin 17 | Baseline, Day 30, 6 months
  Serum Gastrin 17 will be measured and compared to baseline.
Bile acids/salts | Baseline, Day 30
  Bile acids and bile salts can be affected by pH changes. The differential characterization of bile acid and bile salts will be performed at Baseline as compared to Day 30
Serum calcium | Baseline, 30 days and 6 months
Serum magnesium | Baseline, 30 days and 6 months
48 hour gastroesophageal pH measurement | Baseline, 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, M.D., Principal Investigator — Kansas City, Missouri VAMC
Locations (1):
- Veteran's Administration Medical Center, Kansas City, Missouri, United States